CLINICAL TRIAL: NCT05541042
Title: Radiogenomics in Glioblastoma: Correlation Between Multiparametric Imaging Biomarkers and Genetic Biomarkers Based on Tumor Tissues and ctDNA
Brief Title: Radiogenomics in Glioblastoma: Correlation Between Multiparametric Imaging Biomarkers and Genetic Biomarkers
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HPPH-rgGBM
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with glioblastoma
  Interventions: Other: Observational only

INTERVENTIONS:
Other: Observational only — This is an observational study

SUMMARY:
The purpose of this study is to evaluate relationships between multiparametric imaging biomarkers and genetic analysis in glioblastoma patients.

DETAILED DESCRIPTION:
To evaluate relationships between multiparametric imaging biomarkers(CT, PET/CT, MRI) and genetic analysis (tumor tissues and ctDNA in tumor in situ fluid) in glioblastoma patients

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histologically confirmed diagnosis of glioblastoma
* Resection surgery done at the study center (Henan Provincial People's Hospital), with an reservoir intraoperatively implanted connecting the surgical cavity and the subscalp for postoperative noninvasive TISF collection
* Able to tolerable PET/CT and CT imaging required by protocol
* Karnofsky performance status (KPS) of 70 or higher

Exclusion Criteria:

* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring chronic and systemic immunosuppressive treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. Subjects have any other condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalent are permitted in absence of active autoimmune disease
* Clinically significant (i.e., active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment. Any previous venous thromboembolism ≥ NCI CTCAE Grade 3 within 3 months prior to start of study treatment
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study enrollment) use of anticoagulants that, in the opinion of the investigator, would place the subject at significant risk for bleeding.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Functional and genomic profiling of glioblastoma | 3 years after diagnosis
  Prognostic stratification will be evaluated using following parameters:
  Quantitative and qualitative parameters from CT, PET, MRI Genomic data of glioblastoma tumor samples and tumor in situ fluid samples

SECONDARY OUTCOMES:
Relationship between genomic and multiparametric imaging profiling | 3 years after diagnosis
  We will evaluate if certain relationship exists between changes in multiparametric imaging markers from CT, PET, MRI and genomic informations of glioblastoma.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, MD, PhD, Study Director — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No